CLINICAL TRIAL: NCT00100217
Title: Evaluation of Patients With Critical Illness: Intensive Care Training Protocol
Brief Title: Evaluation of Patients With Critical Illness
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050062; 05-CC-0062
Record Dates: First submitted 2004-12-23; First posted 2004-12-24 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-06-25

CONDITIONS: Critical Illness
Keywords: Training; Critical Care; Heart Failure; Pulmonary Hypertension; Infectious Diseases
MeSH Terms: conditions — Critical Illness; Heart Failure; Hypertension, Pulmonary; Communicable Diseases

SUMMARY:
This study provides training opportunities for critical care specialists in evaluating and treating critically ill patients. Patients enrolled in the study receive standard tests and treatments. The study objectives are to:

* Provide additional training for staff of the NIH Clinical Center intensive care unit, including physicians, nurses, fellows, and other trainees so that they develop and maintain essential skills,
* Gather information about the natural history and outcomes of critical illness, accompanying conditions, and complications,
* Develop hypotheses about the medical problems involved in the illnesses and their treatment, and
* Identify critically ill patients who may be eligible for specific NIH research protocols.

Critically ill patients 18 years of age and older who may benefit by transferring to the NIH Clinical Center for treatment may be eligible for this study. Patients will be transferred to the Clinical Center from another hospital only when the referring and accepting physicians in both institutions agree that the potential benefit of coming to the NIH outweighs the risk of transferring the patient.

Participants are evaluated and treated at the Clinical Center. Patients provide a medical history and have a physical examination. They may also have various medical tests and procedures needed to evaluate their condition. These procedures may include blood work, placement of an intravenous (IV) line, x-rays and other imaging tests such as computed tomography (CT) or magnetic resonance imaging (MRI) and other procedures.

Patients who are diagnosed with a specific condition may be offered treatment or may be referred to another study that is more appropriate for that particular problem.

DETAILED DESCRIPTION:
This protocol is designed as a training study, to permit evaluation and treatment of subjects with critical illnesses. A data base, not otherwise obtainable, will be collected of disease processes related to critical illness. Observation of the short-term effects of intensive care interventions will also take place. Minimal studies scheduled for each admission will include a medical history and physical examination, monitoring of hemodynamic status, routine laboratory tests, and evaluation for possible causes of the critical illness. Treatment plans will be individualized for each patient's condition, and the number and length of additional visits and diagnostic evaluations will vary accordingly. Any medical care recommended or provided to the patient will be consistent with routine standards of practice as outlined in Clinical Center (CC) and Critical Care Medicine policies. In selected patients, blood samples may be stored for future research.

The CC is a JCAHO-accredited medical facility with protocols both for standard medical care and also for research. The Critical Care team is made up of intensivists, critical care fellows, nurses, nurse practitioners, and a pharmacist. All of the intensivists are certified in one or more medical subspecialties including critical care and/or cardiology, infectious diseases, pulmonology, and anesthesiology. The CC Medical Intensive Care Unit (MICU) is a state-of-the-art facility that provides comprehensive care for patients with multi-organ failure, sepsis, and medical emergencies. There are daily multi-disciplinary rounds. Attending physicians are in-house during normal business hours and on-call at home at night. A MICU Fellow is always available in-house.

Suitable candidates for this study could include critically ill patients with a diagnostic or therapeutic dilemma, an unusual presentation of disease, or a disease requiring novel therapy available at the CC. Because inter-hospital transfer of the critically ill may increase patient risk, patients will be accepted only if there is a likely medical benefit that outweighs the risk of transfer and if the risk of transfer is thought to be acceptable by both the referring and accepting physicians.

Critically ill patients represent a vulnerable population because of serious illness that may affect their ability to make decisions. They must have an identified durable power of attorney designated for decision making, prior to transfer to the CC.

The risks of this study include the risk of transfer of a critically ill patient from one facility to another and the risks of standard or accepted medical care. There may be no benefit to participation in this study.

In addition to the care available through enrollment in this protocol, patients may also enroll in other NIH protocols if they wish.

The establishment of this protocol will provide a means to evaluate and treat patients, and to generate hypotheses and protocols based on this clinical experience in critical illness.

ELIGIBILITY:
* INCLUSION CRITERIA

Patients are subject to selection by the principal and associate investigators, and will fit any of the following criteria:

Patient with critical illness, who, in the opinion of the accepting physician, may obtain medical benefit by transfer to the CC.

Patient requiring ICU admission according to the SCCM and CCMD guidelines for ICU or intermediate care admissions and with a diagnosis or probable diagnosis on the ICU training protocol diagnosis list or a diagnosis deemed to be appropriate for staff training.

Patient not on the diagnosis list may be admitted at the discretion of the attending physician, if there is prospect of direct medical benefit to the patient.

Age 18 years or older.

Patient may or may not be able to give consent. If the patient is competent, he/she will give written consent prior to transfer to NIH. If the patient is unable to provide informed consent, written witnessed consent will be obtained from the appointed Durable Power of Attorney.

Patient may or may not have other chronic illness.

Patient may be receiving medications for chronic illness treated by their private primary care physicians.

Patient who lacks primary medical care outside the NIH may be enrolled in this protocol, if an appropriate referral can be made to a competent healthcare provider who has agreed to assume care when the patient is discharged.

Patient currently on other NIH protocols requiring ICU admission may be included in this study.

The benefit of transferring the patient to the NIH out weighs the risk of the transfer for the patient.

Available ICU bed in the MICU.

EXCLUSION CRITERIA

Patients with the following problems will be excluded from study:

Patient who does not require critical care.

Patient for whom further therapy is deemed futile by the attending physician.

Patient with known pregnancy, prior to enrollment in the protocol.

Any concurrent condition (medical, social, behavioral), which in the opinion of the medical team would preclude or confound acquisition/interpretation of data or delivery of clinical care.

Less then 18 years of age.

Any patient not requiring ICU admission according to the SCCM and CCMD guidelines for ICU or intermediate care admissions or without a diagnosis or probable diagnosis on the ICU training protocol diagnosis list.

Risk of transfer out weighs the benefit of the transfer for the patient.

No Durable Power of Attorney.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2004-12-21; Study Completion 2010-06-25

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Parrillo JE, Cunnion RE, Epstein SE, Parker MM, Suffredini AF, Brenner M, Schaer GL, Palmeri ST, Cannon RO 3rd, Alling D, et al. A prospective, randomized, controlled trial of prednisone for dilated cardiomyopathy. N Engl J Med. 1989 Oct 19;321(16):1061-8. doi: 10.1056/NEJM198910193211601. PMID 2677721
- [Background] Parker MM, McCarthy KE, Ognibene FP, Parrillo JE. Right ventricular dysfunction and dilatation, similar to left ventricular changes, characterize the cardiac depression of septic shock in humans. Chest. 1990 Jan;97(1):126-31. doi: 10.1378/chest.97.1.126. PMID 2295231
- [Background] Parker MM, Ognibene FP, Parrillo JE. Peak systolic pressure/end-systolic volume ratio, a load-independent measure of ventricular function, is reversibly decreased in human septic shock. Crit Care Med. 1994 Dec;22(12):1955-9. PMID 7988132